CLINICAL TRIAL: NCT05130476
Title: Intraoperative Near-infrared Imaging Techniques for Identifying and Preserving Viable Parathyroid Glands During Total and Completion Thyroidectomy: a Matched Cohort Study
Brief Title: Near-infrared Imaging Techniques for Identifying and Preserving Viable Parathyroid Glands During Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Sanne Høxbroe Michaelsen, Principal investigator, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-20200154
Record Dates: First submitted 2021-11-08; First posted 2021-11-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Hypoparathyroidism Postprocedural
Keywords: Near-infrared fluorescence

STUDY DESIGN:
Intervention Model Description: Matched cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NIRAF+ICGA (Experimental): During thyroid surgery, near-infrared-induced autofluorescence is used for the identification of the parathyroid glands, combined with indocyanine green near-infrared angiography for identification of the parathyroid feeding vessels.
  Interventions: Procedure: Near-infrared-induced autofluorescence and indocyanine green near-infrared angiography

INTERVENTIONS:
Procedure: Near-infrared-induced autofluorescence and indocyanine green near-infrared angiography — During thyroid surgery, near-infrared-induced autofluorescence is used for the identification of the parathyroid glands, combined with indocyanine green near-infrared angiography for identification of the parathyroid feeding vessels.

SUMMARY:
The parathyroid glands and their blood vessels are notoriously difficult to visualize and may therefore be unintentionally and irrevocably damaged during thyroid surgery. This project investigates new surgeon-performed imaging techniques that visualize the parathyroid glands and their vessels in real-time during thyroid surgery. The purpose is to examine, in a matched cohort study, whether the implementation of near-infrared-induced autofluorescence for identification of the parathyroid glands, combined with indocyanine green near-infrared angiography of the parathyroid feeding vessels, can reduce the incidence of postoperative hypocalcaemia in patients undergoing total and completion thyroidectomy at Odense University Hospital.

DETAILED DESCRIPTION:
The most common complication after thyroidectomy is postoperative hypoparathyroidism due to unintentional intraoperative injury, excision, or devascularisation of the parathyroid glands. This complication can be either transient (≤6 months), or permanent (> 6 months). The pooled results from four recent studies from three different Danish university hospitals show that 117/945 patients (12.4%) suffered from permanent hypoparathyroidism after total and completion thyroidectomy. This is a very high percentage, considering that the consequences of hypoparathyroidism and its treatment may be severe and include prolonged hospitalization, neuromuscular symptoms, nephrocalcinosis, nephrolithiasis, premature cataracts, seizures, basal ganglia calcification, and increased mortality.

To minimize the risk of postoperative hypoparathyroidism, the standard approach to thyroidectomy is to keep dissection as close to the thyroid capsule as possible while visually scrutinizing the surgical field for the parathyroid glands and their delicate feeding vessels. In spite of these measures, the reported incidences of transient and permanent hypocalcaemia clearly demonstrate a need to further decrease the risk of inadvertent injury to the parathyroid glands and their vessels during thyroid surgery. To achieve this goal, surgeons need a reliable intraoperative aid that can 1) help them identify the parathyroid glands in vivo and 2) locate their feeding vessels and evaluate their perfusion in real-time during thyroid surgery. Recently, two near-infrared fluorescence techniques have emerged, that could potentially meet the requirement of identifying the parathyroid glands and assessing their vasculature using the same piece of technical equipment. The techniques are: near-infrared-induced autofluorescence of the parathyroid glands (NIRAF) for parathyroid identification, and indocyanine green near-infrared angiography (ICGA) for the assessment of parathyroid vascularization. A recent systematic review concluded that these most reported-on optical tools for parathyroid identification and perfusion assessment are favourable for clinical application in terms of being real-time and non-invasive, having a high sensitivity, an excellent safety profile, and involving no exposure to ionizing radiation. Prior to a broader implementation, commercially unaffiliated investigator-initiated studies are needed to evaluate the clinical effect of the bimodal application of NIRAF and ICGA on the incidence of postoperative hypoparathyroidism after total and completion thyroidectomy. This study intends to address this need.

The hypothesis of the study is that near-infrared-induced autofluorescence (NIRAF) combined with indocyanine green near-infrared angiography (ICGA) of the parathyroid glands can reduce the incidence of permanent hypoparathyroidism after total and completion thyroidectomy to 1/3 or less of the incidence in a matched retrospective control group.

ELIGIBILITY:
Inclusion Criteria:

• Patients 18 years and older who are scheduled to undergo total or completion thyroidectomy at the department of Oro-Rhino-Laryngology (ORL) and Head and Neck Surgery at Odense University Hospital, Denmark.

Exclusion Criteria:

* Not legally competent.
* Does not read or speak Danish.
* Is pregnant or nursing.
* Suffers from chronic kidney disease with an estimated glomerular filtration rate < 45 ml/min/1.73m2.
* Has a history of allergy to iodides or to indocyanine green.
* Suffers from hyperparathyroidism, hypoparathyroidism, or hypocalcaemia prior to surgery.
* Prescription use of supplemental active vitamin D: dihydrotachysterol (ATC 11CC02), alfacalcidol (ATC A11CC03), or calcitriol (ATC A11CC04).
* Patients scheduled to have a radioactive iodine uptake study performed ≤ 7 days after the thyroidectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Permanent hypoparathyroidism 12 months after surgery | 12 months postoperatively
  The number of participants in the study cohort with permanent hypoparathyroidism 12 months after treatment compared to the number of participants with permanent hypoparathyroidism 12 months after treatment in a matched retrospective cohort from the same hospital that underwent surgery without NIRAF+ICGA.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://open.rsyd.dk/OpenProjects/openProject.jsp?openNo=1434&lang=da